CLINICAL TRIAL: NCT04325776
Title: A Randomized, Double-blind and Imitation, Parallel-control, Multicenter Phase II Study of AL2846 Versus Zoledronic Acid in Subjects With Advanced Non-small Cell Lung Cancer (NSCLC) With Bone Metastasis
Brief Title: A Study of AL2846 Versus Zoledronic Acid in Subjects With Advanced Non-Small Cell Lung Cancer With Bone Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL2846-II-01
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-03

CONDITIONS: Bone Metastatic Non-small Cell Lung Cancer
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL2846+An analog of zoledronic acid injection (Experimental): AL2846 capsules 150 mg given orally, once daily in 28-day cycle, an analog of zoledronic acid injection (5ml:0mg) administered intravenously (IV) on Day 1 of each 28-day cycle.
  Interventions: Drug: AL2846
- An analog of AL2846+ zoledronic acid injection (Active Comparator): An analog of AL2846 capsules 0 mg given orally, once daily in 28-day cycle, zoledronic acid injection (5ml:4mg) administered intravenously (IV) on Day 1 of each 28-day cycle.
  Interventions: Drug: Zoledronic Acid Injection

INTERVENTIONS:
Drug: AL2846 — AL2846 is a multi-target tyrosine kinase receptor inhibitor with obvious selective to c-met.
  Arms: AL2846+An analog of zoledronic acid injection
Drug: Zoledronic Acid Injection — Zoledronic acid is a bisphosphonate drug that has a strong inhibition of bone resorption and a potential to promote bone formation, and can be used for bone metastasis caused by malignant tumors.
  Arms: An analog of AL2846+ zoledronic acid injection

SUMMARY:
AL2846 is a multi-target tyrosine kinase receptor inhibitor with obvious selective to c-met, suggesting that its anti-tumor effect mainly inhibits the activation of key downstream oncogenic pathways by inhibiting expression of c-met, tumor angiogenesis and tumor cell migration.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form. 2.18 years and older; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

  3.Histologically confirmed advanced non-small cell lung cancer with at least one bone metastatic lesion with bone destruction.

  4.Has received at least two systematic treatment regimens that failed or were unable to tolerate treatment.

  5.EGFR, ALK gene mutations are negative. 6.Adequate laboratory indicators. 7.No pregnant or breastfeeding women, and a negative pregnancy test.

Exclusion Criteria:

* 1.Small cell lung cancer. 2. Diagnosed and/or treated additional malignancy within 5 years with the exception of cured cervical carcinoma in situ and non-melanoma skin cancer.

  3. Has received radiotherapy, chemotherapy and surgery before and less than 4 weeks from the first administration and less than 5 half-lives of oral targeted drugs after the completion of treatment.

  4. Has received systemic radionuclide therapy or semi-extracorporeal radiation for bone metastases.

  5. Has known to be allergic to the study drug or any of its excipients. 6. Has symptomatic brain metastases, spinal cord compression, and cancerous meningitis within 8 weeks,or brain or pia mater disease confirmed by CT or MRI examination before the first dose.

  7. Has adverse events caused by previous therapy that did not recover to ≤ grade 1, with the exception of alopecia or ≥ grade 2 neurotoxicity caused by Oxaliplatin.

  8. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear.

  9. Has spinal cord compression or mandibular osteonecrosis. 10.Has multiple factors that affect oral medications. 11.Has gastroduodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases or other conditions judged by the investigator that may cause gastrointestinal bleeding or perforation.

  12.Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

  13. Has severe acute comorbidities before the first dose. 14. Has participated in other clinical trials within 4 weeks before the first dose.

  15.According to the investigators' judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The time when the first bone-related event (SRE) occurred | up to 96 weeks
  The time from the randomization to the first occurrence of any meeting of bone-related event criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 96 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause, based on investigator.
Overall response rate (ORR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Effectiveness of improving average daily pain intensity on week 8 and 16 (Refer to Brief pain inventory (BPI) and the Verbal rating scale (VRS) | on 8 and 16 week
  Referring to Brief pain inventory (BPI) and Verbal rating scale (VRS), the percentage of improvement in the average intensity of pain confirmed at week 8 and week 16 compared to the previous average intensity.
Biomarkers | up to 96 weeks
  Relationship between drug efficacy and related biomarkers such as C-Met, FGFR, c-Kit, RET.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Anhui Chest Hospital, Hefei, Anhui
  - Henan Cancer Hospital, Zhengzhou, Henan
  - China-Japan Union Hospital Of Jilin University, Changchun, Jilin
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - Shenyang Chest Hospital, Shenyang, Liaoning
  - Sir Run Run Shaw Hospital (SRRSH), Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang